CLINICAL TRIAL: NCT03894228
Title: Safety of IBD Drugs During Pregnancy and Breastfeeding: Mothers and Babies' Outcomes (DUMBO Registry)
Status: Recruiting | Type: Observational
Sponsor: Grupo Espanol de Trabajo en Enfermedad de Crohn y Colitis Ulcerosa (Other)
Collaborators: Spanish Agency of Medicines and Health Products (Other Government)
Responsible Party: Sponsor
Other Study IDs: GIS-DUMBO-2018
Record Dates: First submitted 2018-12-17; First posted 2019-03-28 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Inflammatory Bowel Diseases; Pregnancy
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 57 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Biologics exposed cohort: Children born from mothers treated with biologic drugs (with or without immunomodulators) at any time during pregnancy or the three months before conception. Biologic drugs are IgG monoclonal antibodies able to cross the placenta.
- Immunomodulators exposed cohort: Children born from mothers treated with immunomodulators (without biologics) during pregnancy or the three months before conception.
- Non-exposed cohort: Children born from mothers treated neither with biologic drugs nor with immunomodulators at any time during pregnancy or the three months before conception.

SUMMARY:
This is a prospective, observational, multicenter registry, which will enrol pregnant women with IBD (CD, UC, or unclassified IBD) over 5 years in Spain.

In addition, each incident gestation will be followed-up during pregnancy, and children born to those mothers will be followed-up over 4 years to determine the incidence of serious adverse events (such as alteration of developmental status, infections, neoplasia or any other serious adverse events) during the study period. In order to harmonize the inclusion of adverse events and complications, only serious adverse events will be registered . The main variable will be the development of serious infection in children as this is the outcome that had controversial results in previous studies.

DETAILED DESCRIPTION:
OBJECTIVES Main objective - To assess the safety of drugs used for IBD treatment both for pregnancy and for the offspring mainly focused on the risk of serious infections (from birth and in the first 4 years of life).

Specific objectives

* To know the risk of serious adverse events (including abortions) during pregnancy and delivery associated with drugs used for the treatment of IBD.
* To asses the developmental status of children born from IBD mothers during the first 4 years.
* To compare the relative risk of serious adverse events in children born from mothers with IBD who have been exposed in utero to different drugs to treat IBD with the risk in children who were not exposed.
* To compare the prevalence of malformations in children exposed to drugs to treat IBD in utero with the prevalence in children who were not exposed.
* To evaluate the relative risk of developing neoplasm in children exposed to drugs to treat IBD.

Inclusion criteria

* Patients over 18 years of age diagnosed with IBD.
* Confirmed pregnancy.
* Awareness of the pregnancy (by the researcher) before week 28th of gestation (the end of the second trimester).

Exclusion criteria. - Patients who do not accept to participate in the study Study cohorts

- Biologics exposed cohort: Children born from mothers treated with biologic drugs (with or without immunomodulators) at any time during pregnancy or the three months before conception. Biologic drugs are IgG monoclonal antibodies able to cross the placenta.

* Immunomodulators exposed cohort: Children born from mothers treated with immunomodulators (without biologics) during pregnancy or the three months before conception.
* Non-exposed cohort: Children born from mothers treated neither with biologic drugs nor with immunomodulators at any time during pregnancy or the three months before conception.

Tasks and responsibilities:

IBD specialists from the participating centers will be responsible for identifying the patients, obtaining the informed consent and registering them in the database.

Each participating investigator will register all the demographic and clinical data of the mother at the time of entering in the study and will contact the pregnant woman at the end of first trimester, the end of second trimester, the end of third trimester and one month after delivery to prospectively include information about disease activity, treatments and serious adverse events (if any) during pregnancy and delivery. If the mother contacts the clinician (researcher) after the end of the first trimester but before the end of the second trimester of gestation, the case can be included and data up to the entry date registered retrospectively. In order to ensure data quality, patients who inform about the pregnancy after the end of the second trimester of gestation will be excluded.

After birth, the mother will be contacted every 3 months to include information about the child development and serious adverse events (mainly malformations, infections, hospital admissions or neoplasias such as developmental tumors). After consenting, contact information of the mother will be shared with the research team in Hospital Universitario de La Princesa in order to complete the information every 3 months. On a yearly basis, the mothers will provide the site investigator with the reports that support the information given in the remote contact. In addition, in the first visit after birth, mothers will be provided with the Ages and Stages Questionnaire (ASQ 3, annex 2) that should be completed during follow-up (2, 4, 6, 8, 9, 10, 12, 14, 16, 18, 20, 22, 24, 27, 30, 33, 36, 42, 48 months of age). The mother should give the questionnaire she has completed once per year. External monitoring of cases included in the registry will also be performed by review of some cases selected at random by the research team of Hospital Universitario de La Princesa.

Definitions

1. Disease location and phenotype: IBD location and phenotype will be defined according to the Montreal classification.
2. Date of conception: It will be defined as the date of last menstruation before becoming pregnant.
3. Smoking: Smoking status will be categorized as "non-smoker", "smoker", or "ex-smoker", and will be considered at the time of conception. Patients will be considered "smokers" if they smoked more than 7 cigarettes per week for at least 6 months prior to conception. Patients will be considered "ex-smokers" if they quit smoking before conception. Patients will be considered "non-smokers" if they never smoked.

3. Diagnosis of pregnancy: Elevated human chorionic gonadotropin (hCG) hormone in blood or urine (biochemical pregnancy).

4. Miscarriage: Natural death of an embryo or fetus before it is able to survive independently.

5. Elective abortion: The removal of an embryo or fetus from the uterus in order to end a pregnancy.

6. Comorbidities: Mother's diseases, with special mention to hypertension, diabetes mellitus, seizure disorders, thyroid disorders, allergic disorders, heart diseases, connective tissue diseases, autoimmune diseases, hepatitis.

7. Known risk factors for adverse pregnancy outcomes, including environmental or occupational exposure, among others.

8. Treatments: Treatments received by the mother in the 3 months before conception, during pregnancy and breastfeeding will be recorded.

9. Serious adverse events: In order to harmonize the inclusion of adverse events and complications, only serious adverse events will be registered (see the definition of adverse events in the Annex 1 of the protocol). Nevertheless, the investigators have predefined the most frequent serious adverse events during pregnancy and in the offspring. In this respect, the main variable in our study will be the development of serious infection in the offspring (infection meeting criteria of serious adverse event).

9.1. Serious adverse events during pregnancy: Any event that meets the criteria of serious adverse event will be registered in the database. Some of the most frequent serious adverse events during pregnancy are specifically defined and inquired by the registry: abortion, stillbirth, growth retardation, serious infection, eclampsia, placenta previa, chorioamnionitis, or abruptio placenta. Abnormalities found in the 20th week ultrasound will be registered (although malformations should be confirmed after birth and included in the Serious Adverse Events section of the newborn). Fetal malformations that lead to abortion or stillbirth will be included as cause of abortion or cause of stillbirth in their specific sections (Serious adverse events of the mother).

9.2. Serious adverse events during delivery: Serious adverse events, such as instrumental delivery or preterm delivery will be registered in the Serious adverse events of the mother section. The admission for delivery will not be considered as a serious adverse event, but any event causing prolongation of the admission will be considered as a serious adverse event and registered in the specific section.

9.3. Serious adverse events in the newborns and children: Serious adverse events in the newborn and children, such as congenital malformations, admission to the intensive care unit, low birth weight, hypoxic-ischemic encephalopathy, neonatal stroke or low Apgar score, severe infections and tumors will be included.

10. Preterm delivery: Delivery before week 37 of gestation18, 19. 11. Low birth weight: <2,500 mg18, 19. 12. IBD activity: The IBD activity will be assessed at conception (when the physician is aware of the pregnancy) and in each trimester of gestation based on the Harvey-Bradshaw for CD and Partial Mayo Score for UC patients.

13. Low Apgar score: Apgar scores lower than 7 are considered low, and scores of 7 or higher are considered normal at ten minutes after birth20.

14. Serious infection: Only infections that meet the criteria of serious adverse event will be included. The inclusion of any infection, irrespective of its seriousness, would be very heterogeneous among investigators, leading to reporting bias which might affect the interpretation of the results. This variable will be the main outcome.

15. Developmental status: The developmental status will be assessed by the ASQ-3 questionnaire (annex 2). The mothers will complete the questionnaire at home and send the completed forms yearly to their treating clinicians.

Data collection and follow-up After the case is registered, four other visits will be recorded during pregnancy, coinciding with the routine visits of the patient for the follow-up of her disease. After delivery, the children will be followed-up until the age of 4 years. In case of multiple gestations, each child will be considered as a case with his/her own follow-up. Only live newborns will be considered cases. Abortions or stillbirths will be registered as mothers' adverse events. In multiple gestations, the number of fetuses affected by a certain serious adverse event will be indicated in the CRF. During the child's follow-up period, the mother (that is the patient, indeed) will be contacted remotely every-three months to complete information about child complications (if any). The visits over the study are described below. The variables included in the eCRF are listed in Annex 3.

* Visit 0 (baseline): inclusion of patient in the study (after confirmed pregnancy) and registration of clinical data (characteristics of the disease, disease activity and treatments).
* Visit 1 (end of first trimester of gestation): Updating of data related to treatment, disease activity and serious adverse events (if any).
* Visit 2 (end of second trimester of gestation): Updating of data related to treatment, disease activity and serious adverse events (if any).
* Visit 3 (end of third trimester of gestation): Updating of data related to treatment, disease activity and serious adverse events (if any).
* Visit 4 (1 month after delivery): Updating of data related to treatment, disease activity and serious adverse events (if any). In addition, in this visit, the child will be registered in the database as a case. Information of the newborn, such as date of birth, sex, birth weight, Apgar score (at 5 and 10 minutes), vaccines, breastfeeding, serious adverse events, etc., will be included.
* Visit 5 (3 months of age, 2 months after visit 4) to 20 (4 years of age): Updating of data related to children development, vaccines, breastfeeding, date of schooling, infections, hospitalizations, allergies or any other complications. The same data will be queried to the mother every-three months after the age of 4 years. Remote contacts will be allowed to complete the children information, as the investigators believe that this way of obtaining information will not have impact on the quality of data and will improve the adherence to the protocol. Nevertheless, once per year data should be confirmed with medical reports provided by the mothers.

Study data will be collected and managed using an electronic data capture tool (Research Electronic Data Capture [REDCap]1, 18, 19), which is hosted at Asociación Española de Gastroenterología21, a non-profit scientific and medical society focusing on gastroenterology. AEG provides this service free of charge, with the sole aim of promoting independent investigator-driven research. REDCap is a secure, web-based application designed to support data capture for research studies that provides the following: 1) an intuitive interface for validated data entry; 2) audit trails for tracking data manipulation and export procedures; 3) automated export procedures for seamless data downloads to common statistical packages; and 4) procedures for importing data from external sources.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age diagnosed with IBD.
* Confirmed pregnancy.
* Awareness of the pregnancy (by the researcher) before week 28th of gestation (the end of the second trimester).

Exclusion Criteria:

• Patients who do not accept to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women.
Study Population: Pregnant women with IBD (CD, UC, or unclassified IBD) over 5 years in Spain.
Sampling Method: Probability Sample
Enrollment: 1750 (Estimated)
Dates: Start 2019-05-21 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
To calculate the incide rate of serious infections during pregnancy (evaluated and the end of pregnancy) based on the medications used to treat IBD. | 9 months
  To assess the prevalence of complications related to drugs used for IBD treatment for pregnancy.
To calculate the incide rate of serious infections for the offspring (at eh age of 4 years) based on the medications used to treat IBD. | 4 years
  To assess the prevalence of complications related to drugs used for IBD treatment for the offspring.
To calculate the incide rate of serious adverse events during pregnancy (evaluated at the end of pregnancy) based on the medications used to treat IBD. | 9 months
  To asses the prevalence of complications related to drugs used for IBD treatment for pregnancy.
To calculate the incide rate of serious adverse events during offspring (at the age of 4 years) based on the medications used to treat IBD. | 4 years
  To asses the prevalence of complications related to drugs used for IBD treatment for offspring mainly focused on the risck of serious infections at the age of 4 years.

SECONDARY OUTCOMES:
2. To calculate the Odds ratio of serious adverse events (including abortions) during pregnancy and delivery based on the drugs used for the treatment of IBD. | 4 years and 9 months
  To know the risk of serious adverse events (including abortions) during pregnancy and delivery associated with drugs used for the treatment of IBD.
3. To measure the developmental status of children born from IBD mothers with the ASQ-3 questionnaire during the first 4 years. | 4 years and 9 months
  To asses the developmental status of children born from IBD mothers during the first 4 years.
4. To calculate the Hazard ratio of serious adverse events in children born from mothers with IBD who have been exposed in utero to different drugs to treat IBD with the risk in children who were not exposed. | 4 years and 9 months
  To compare the relative risk of serious adverse events in children born from mothers with IBD who have been exposed in utero to different drugs to treat IBD with the risk in children who were not exposed.
5. To calculate the proportion of children with malformations and to compare the proportions between exposure groups (children exposed to biologics with those non exposed to these drugs). | 4 years and 9 months
  To compare the prevalence of malformations in children exposed to biologics to treat IBD in utero with the prevalence in children who were not exposed
6. To calculate the Hazard ratio of developing neoplasm in children exposed to drugs to treat IBD. | 4 years and 9 months
  To evaluate the relative risk of developing neoplasm in children exposed to drugs to treat IBD.

CONTACTS AND LOCATIONS:
Locations (73):
- Spain (73):
  - Complejo Hospitalario Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital Universitario Reina Sofía, Córdoba, Andalusia
  - Hospital Clínico Universitario San Cecilio, Granada, Andalusia
  - Hospital Infanta Elena, Huelva, Andalusia
  - Hospital Universitario Juan Ramón Jimenez, Huelva, Andalusia
  - Hospital Regional Universitario de Málaga, Málaga, Andalusia
  - Hospital Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital San Juan de Dios del Aljarafe, Seville, Andalusia
  - Hospital Universitario Virgen del Rocío, Seville, Andalusia
  - Hospital San Jorge, Huesca, Aragon
  - Hopsital Universitario Miguel Servet, Zaragoza, Aragon
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza, Aragon
  - Hospital Royo Villanova, Zaragoza, Aragon
  - Hospital Comaral de Inca, Palma de Mallorca, Balearic Islands
  - Hospital Universitario de Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario de Álava, Alava, Basque Country
  - Hospital Universitario de Donostia, Donostia / San Sebastian, Basque Country
  - Hospital de Galdakao-Usansolo, Galdakao, Basque Country
  - Hospital Doctor Negrin, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - Hospital Universitario Nuestra Señora de la Candelaria, Santa Cruz de Tenerife, Canary Islands
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital General de Castellon, Castellon, Castellón
  - Hospital Santos Reyes, Burgos, Castille and León
  - Hospital Universitario de Burgos, Burgos, Castille and León
  - Hospital Universitario de Salamanca, Salamanca, Castille and León
  - Hospital Clínico de Valladolid, Valladolid, Castille and León
  - Hospital Provincial de Zamora, Zamora, Castille and León
  - Hospital Virgen de la Concha, Zamora, Castille and León
  - Hospital Alcázar de San Juan, Ciudad Real, Castille-La Mancha
  - Hospital General de Tomelloso, Ciudad Real, Castille-La Mancha
  - Hospital General Universitario de Ciudad Real, Ciudad Real, Castille-La Mancha
  - Hospital Virgen de la Salud, Toledo, Castille-La Mancha
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Universitario Clinic i Provincial, Barcelona, Catalonia
  - Hospital Universitario de Bellvitge, Barcelona, Catalonia
  - Hospital Vall d´Hebron, Barcelona, Catalonia
  - Hospital Universitari Dr Josep Trueta, Girona, Catalonia
  - Hospital Sant Joan de Déu, Manresa, Catalonia
  - Consorci Sanitari de Terrassa, Tarragona, Catalonia
  - Hospital Joan XXIII, Tarragona, Catalonia
  - Hospital Universitari Sant Joan de Reus, Tarragona, Catalonia
  - Hospital San Pedro Alcántara, Cáceres, Extremadura
  - Complexo Hospitalario Universitario de A Coruña, A Coruña, Galicia
  - Complejo Hospitalario Universitario de Ferrol, Ferrol, Galicia
  - Complexo Hospitalario Universitario de Ourense, Ourense, Galicia
  - Hospital Alvaro Cunqueiro, Vigo, Galicia
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hosptial Universitario Infanta Cristina, Parla, Madrid
  - Hospital del Henares, San Fernando de Henares, Madrid
  - Hospital Universitario de Torrejón, Torrejón, Madrid
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital General Universitario de Alicante, Alicante, Valencia
  - Hospital Marina Baixa de Villajoyosa, Alicante, Valencia
  - Hospital Universitario San Juan, Alicante, Valencia
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Lluis Alcanyís de Xátiva, Valencia, Valencia
  - Hospital Universitàri i Politècnic La Fe, Valencia, Valencia
  - Hospital de Granollers, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario de La Paz, Madrid
  - Hospital Universitario Doce de Octubre, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Infanta Sofía, Madrid
  - Hospital Universitario Rey Juan Carlos, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Virgen del Rosell, Murcia
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gisbert JP. Safety of immunomodulators and biologics for the treatment of inflammatory bowel disease during pregnancy and breast-feeding. Inflamm Bowel Dis. 2010 May;16(5):881-95. doi: 10.1002/ibd.21154. PMID 19885906
- [Background] Gisbert JP, Chaparro M. Safety of anti-TNF agents during pregnancy and breastfeeding in women with inflammatory bowel disease. Am J Gastroenterol. 2013 Sep;108(9):1426-38. doi: 10.1038/ajg.2013.171. Epub 2013 Jun 11. PMID 23752881
- [Background] Burisch J, Pedersen N, Cukovic-Cavka S, Turk N, Kaimakliotis I, Duricova D, Shonova O, Vind I, Avnstrom S, Thorsgaard N, Krabbe S, Andersen V, Dahlerup Jens F, Kjeldsen J, Salupere R, Olsen J, Nielsen KR, Manninen P, Collin P, Katsanos KH, Tsianos EV, Ladefoged K, Lakatos L, Bailey Y, O'Morain C, Schwartz D, Odes S, Martinato M, Lombardini S, Jonaitis L, Kupcinskas L, Turcan S, Barros L, Magro F, Lazar D, Goldis A, Nikulina I, Belousova E, Fernandez A, Hernandez V, Almer S, Zhulina Y, Halfvarson J, Tsai HH, Sebastian S, Lakatos PL, Langholz E, Munkholm P; EpiCom Group. Initial disease course and treatment in an inflammatory bowel disease inception cohort in Europe: the ECCO-EpiCom cohort. Inflamm Bowel Dis. 2014 Jan;20(1):36-46. doi: 10.1097/01.MIB.0000436277.13917.c4. PMID 24252978
- [Background] Mix E, Goertsches R, Zett UK. Immunoglobulins--basic considerations. J Neurol. 2006 Sep;253 Suppl 5:V9-17. doi: 10.1007/s00415-006-5002-2. PMID 16998762
- [Background] Israel EJ, Simister N, Freiberg E, Caplan A, Walker WA. Immunoglobulin G binding sites on the human foetal intestine: a possible mechanism for the passive transfer of immunity from mother to infant. Immunology. 1993 May;79(1):77-81. PMID 8509144
- [Background] Chaparro M, Gisbert JP. Transplacental transfer of immunosuppressants and biologics used for the treatment of inflammatory bowel disease. Curr Pharm Biotechnol. 2011 May;12(5):765-73. doi: 10.2174/138920111795470903. PMID 21342120
- [Background] Julsgaard M, Christensen LA, Gibson PR, Gearry RB, Fallingborg J, Hvas CL, Bibby BM, Uldbjerg N, Connell WR, Rosella O, Grosen A, Brown SJ, Kjeldsen J, Wildt S, Svenningsen L, Sparrow MP, Walsh A, Connor SJ, Radford-Smith G, Lawrance IC, Andrews JM, Ellard K, Bell SJ. Concentrations of Adalimumab and Infliximab in Mothers and Newborns, and Effects on Infection. Gastroenterology. 2016 Jul;151(1):110-9. doi: 10.1053/j.gastro.2016.04.002. Epub 2016 Apr 8. PMID 27063728
- [Background] Vermeire S, Carbonnel F, Coulie PG, Geenen V, Hazes JM, Masson PL, De Keyser F, Louis E. Management of inflammatory bowel disease in pregnancy. J Crohns Colitis. 2012 Sep;6(8):811-23. doi: 10.1016/j.crohns.2012.04.009. Epub 2012 May 16. PMID 22595185
- [Background] Chaparro M, Verreth A, Lobaton T, Gravito-Soares E, Julsgaard M, Savarino E, Magro F, Biron AI, Lopez-Serrano P, Casanova MJ, Gompertz M, Vitor S, Arroyo M, Pugliese D, Zabana Y, Vicente R, Aguas M, Shitrit BA, Gutierrez A, Doherty GA, Fernandez-Salazar L, Cadilla MJ, Huguet JM, O'Toole A, Stasi E, Marcos MN, Villoria A, Karmiris K, Rahier JF, Rodriguez C, Palomares DM, Fiorino G, Benitez JM, Principi M, Naftali T, Taxonera C, Mantzaris G, Sebkova L, Iade B, Lissner D, Bradley FI, Roman LA, Marin-Jimenez I, Merino O, Sierra M, Van Domselaar M, Caprioli F, Guerra I, Peixe P, Piqueras M, Rodriguez-Lago I, Ber Y, van Hoeve K, Torres P, Gravito-Soares M, Rudbeck-Resdal D, Bartolo O, Peixoto A, Martin G, Armuzzi A, Garre A, Donday MG, de Carpi MFJ, Gisbert JP. Long-Term Safety of In Utero Exposure to Anti-TNFalpha Drugs for the Treatment of Inflammatory Bowel Disease: Results from the Multicenter European TEDDY Study. Am J Gastroenterol. 2018 Mar;113(3):396-403. doi: 10.1038/ajg.2017.501. Epub 2018 Feb 20. PMID 29460920
- [Background] Domenech E, Gisbert JP. Efficacy and safety of vedolizumab in the treatment of ulcerative colitis. Gastroenterol Hepatol. 2016 Dec;39(10):677-686. doi: 10.1016/j.gastrohep.2015.11.010. Epub 2016 Mar 2. English, Spanish. PMID 26948838
- [Background] Gisbert JP, Domenech E. [Vedolizumab in the treatment of Crohn's disease]. Gastroenterol Hepatol. 2015 May;38(5):338-48. doi: 10.1016/j.gastrohep.2014.12.003. Epub 2015 Jan 23. Spanish. PMID 25619903
- [Background] Beaulieu DB, Ananthakrishnan AN, Martin C, Cohen RD, Kane SV, Mahadevan U. Use of Biologic Therapy by Pregnant Women With Inflammatory Bowel Disease Does Not Affect Infant Response to Vaccines. Clin Gastroenterol Hepatol. 2018 Jan;16(1):99-105. doi: 10.1016/j.cgh.2017.08.041. Epub 2017 Sep 1. PMID 28870657
- [Background] Lahat A, Shitrit AB, Naftali T, Milgrom Y, Elyakim R, Goldin E, Levhar N, Selinger L, Zuker T, Fudim E, Picard O, Yavzori M, Ben-Horin S. Vedolizumab Levels in Breast Milk of Nursing Mothers With Inflammatory Bowel Disease. J Crohns Colitis. 2018 Jan 5;12(1):120-123. doi: 10.1093/ecco-jcc/jjx120. PMID 28961712
- [Background] Julsgaard M, Kjeldsen J, Bibby BM, Brock B, Baumgart DC. Vedolizumab Concentrations in the Breast Milk of Nursing Mothers With Inflammatory Bowel Disease. Gastroenterology. 2018 Feb;154(3):752-754.e1. doi: 10.1053/j.gastro.2017.08.067. Epub 2017 Oct 5. No abstract available. PMID 28988916
- [Background] Mahadevan U, Vermeire S, Lasch K, Abhyankar B, Bhayat F, Blake A, Dubinsky M. Vedolizumab exposure in pregnancy: outcomes from clinical studies in inflammatory bowel disease. Aliment Pharmacol Ther. 2017 Apr;45(7):941-950. doi: 10.1111/apt.13960. Epub 2017 Feb 7. PMID 28169436
- [Background] Gisbert JP, Chaparro M. Ustekinumab to treat Crohn's disease. Gastroenterol Hepatol. 2017 Dec;40(10):688-698. doi: 10.1016/j.gastrohep.2017.08.006. Epub 2017 Oct 16. English, Spanish. PMID 29042094
- [Background] Rowan CR, Cullen G, Mulcahy HE, Keegan D, Byrne K, Murphy DJ, Sheridan J, Doherty GA. Ustekinumab Drug Levels in Maternal and Cord Blood in a Woman With Crohn's Disease Treated Until 33 Weeks of Gestation. J Crohns Colitis. 2018 Feb 28;12(3):376-378. doi: 10.1093/ecco-jcc/jjx141. PMID 29045603
- [Background] Nguyen GC, Seow CH, Maxwell C, Huang V, Leung Y, Jones J, Leontiadis GI, Tse F, Mahadevan U, van der Woude CJ; IBD in Pregnancy Consensus Group; Canadian Association of Gastroenterology. The Toronto Consensus Statements for the Management of Inflammatory Bowel Disease in Pregnancy. Gastroenterology. 2016 Mar;150(3):734-757.e1. doi: 10.1053/j.gastro.2015.12.003. Epub 2015 Dec 11. PMID 26688268
- [Background] van der Woude CJ, Ardizzone S, Bengtson MB, Fiorino G, Fraser G, Katsanos K, Kolacek S, Juillerat P, Mulders AG, Pedersen N, Selinger C, Sebastian S, Sturm A, Zelinkova Z, Magro F; European Crohn's and Colitis Organization. The second European evidenced-based consensus on reproduction and pregnancy in inflammatory bowel disease. J Crohns Colitis. 2015 Feb;9(2):107-24. doi: 10.1093/ecco-jcc/jju006. PMID 25602023
- [Background] Boyd HA, Basit S, Harpsoe MC, Wohlfahrt J, Jess T. Inflammatory Bowel Disease and Risk of Adverse Pregnancy Outcomes. PLoS One. 2015 Jun 17;10(6):e0129567. doi: 10.1371/journal.pone.0129567. eCollection 2015. PMID 26083614
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Derived] Palomino L, Velasco Rodriguez-Belvis M, Casanova MJ, Leo-Carnerero E, Calvino-Suarez C, Rivero M, Calvo M, Arroyo MT, Fernandez-Clotet A, Perez-Martinez I, Masedo Gonzalez A, Hernandez V, Ruiz-Cerulla A, Lopez Serrano P, Vega P, Rodriguez-Lago I, Lidon RV, De Jorge MA, Guerra I, Garcia LA, Molina Arriero G, Hervias Cruz D, Busquets D, Gutierrez Casbas A, Van Domselaar M, Valldosera Gomis G, Vazquez Moron JM, Piqueras Cano M, Lucendo AJ, Martin Arranz MD, Ramirez de la Piscina P, Martinez Tirado MDP, Robles Alonso V, Marin Pedrosa S, Camargo Camero R, Armesto Gonzalez E, Tardillo Marin C, Bernardos Martin E, Rodriguez Grau MC, Huguet JM, Marquez-Mosquera L, Sendra Rumbeu P, Bujanda L, Castano-Milla C, Sainz Arnau E, Hernandez L, Ramos L, Bosca-Watts MM, Mancenido Marcos N, Sans M, Morales VJ, Acosta D, Garre A, Munoz Codoceo R, Garcia-Salido A, Gisbert JP, Chaparro M; DUMBO study group of GETECCU. Psychomotor Development in Infants Following Maternal Exposure to Biologics: Results From the DUMBO Registry. Clin Gastroenterol Hepatol. 2025 Jun 13:S1542-3565(25)00488-4. doi: 10.1016/j.cgh.2025.05.012. Online ahead of print. PMID 40518059
- [Derived] Chaparro M, Donday MG, Abad-Santos F, Martin de Carpi FJ, Macia-Martinez MA, Montero D, Acosta D, Brenes Y, Gisbert JP. The safety of drugs for inflammatory bowel disease during pregnancy and breastfeeding: the DUMBO registry study protocol of GETECCU. Therap Adv Gastroenterol. 2021 Jun 3;14:17562848211018097. doi: 10.1177/17562848211018097. eCollection 2021. PMID 34158835

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT03894228/Prot_SAP_000.pdf